CLINICAL TRIAL: NCT04179578
Title: The Value of Lateral Release in Reconstruction of the Diaphragmatic Hiatus in Patients With Type II-IV Paraesophageal Hernia. A Double Blind Randomized Study
Brief Title: The Value of Lateral Release in Reconstruction of the Diaphragmatic Hiatus Hernia
Acronym: PEH2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-02801
Record Dates: First submitted 2019-11-07; First posted 2019-11-27 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Paraesophageal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: Crura plastic or crura plastic with the addition of "lateral release"
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization process is initiated after general anesthesia is induced and the group affiliation will be determined by opening of a sealed envelope specifying the group assignment. The information of group allocation is stored in a closed envelope kept in a locked archive until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crura (Active Comparator): Closure of the diaphragmatic hiatus by a running suture alone
  Interventions: Procedure: Crura plastic
- Crura and lateral release (Active Comparator): Closure of the diaphragmatic hiatus by a running suture and an incision of 4 cm of the left diaphragm (lateral release)
  Interventions: Procedure: Crura plastic

INTERVENTIONS:
Procedure: Crura plastic — Closure of hiatus with a running suture

SUMMARY:
Patients scheduled for surgery for primary paraesophageal herniation are randomized to either conventional suturing of the crura or with the addition of lateral release.

DETAILED DESCRIPTION:
Patient undergoing surgery for primary paraesophageal herniation, are randomized to either conventional suturing of the diaphragmatic crura only or with the addition of a diaphragmatic incision "lateral release".

The patients are examined by computed tomography before surgery and at 1 and 3 years after surgery.

SF-36 (global quality of Life instrument), GSRS (Gastrointestinal Symptoms Rating Scale), Reflux frequency issues and Watson's dysphagia score are completed before and at 3 and 6 month as well as 1 and 3 years after surgery.

Patients undergoing laparoscopic repair for paraesophageal hernia Type II-IV are eligible for inclusion in the study. Included patients will be randomized to either reconstruction of the hiatus by suturing of the crura alone or in combination with an approximately 4 cm incision of the anterior aspect of the left diaphragma "lateral release" before crural suturing. The incision will be covered with a synthetic patch after crural closure is finished. All other aspects of the surgical procedure are similar in the two groups including complete mobilization of the hernia sac before and a total fundoplication after hiatal restoration, respectively.

ELIGIBILITY:
Inclusion Criteria:

* all patients with primary hiatus hernia type II-IV who are deemed suitable for surgery

Exclusion Criteria:

* inability to understand the nature of the purpose of the study and/or to give informed consent.
* American Society of Anesthesiologists physical status-system (ASA) >III
* Achalasia or another severe esophageal motor disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rat of reherniating | 1 year
  computer tomography of abdomen and thorax

SECONDARY OUTCOMES:
complications after operation | 1 year
  symptomatic recurrence
change in quality of life | 1 year
  SF-36 (Quality of Life issues) The SF-36 It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. Higher scores mean a better outcome.
Patients analgesic consumption after operation | 1 year
  information from the patient and the patient´s journal
Length of Stay (LOS) | 1 year
  Information from the patient's journal
sick leave period | 1 year
  Days, information from the patient
GSRS Gastrointestinal Symptom Rating Scale | 1 year
  Scoring;The questionnaire, which contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
  A mean value for the items in each dimension should be calculated:
  Diarrhoea syndrome: 11. Increased passage of stools 12. Loose stools 14. Urgent need for defecation Indigestion syndrome: 6. Borborygmus 7. Abdominal distension 8. Eructation 9. Increased flatus Constipation syndrome: 10. Decreased passage of stools 13. Hard stools 15. Feeling of incomplete evacuation Abdominal pain syndrome: 1. Abdominal pain 4. Sucking sensations 5. Nausea and vomiting Reflux syndrome: 2. Heartburn 3. Acid regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsoposidis A, Thorell A, Axelsson H, Reuterwall Hansson M, Lundell L, Wallenius V, Kostic S, Hakanson B. The value of "diaphragmatic relaxing incision" for the durability of the crural repair in patients with paraesophageal hernia: a double blind randomized clinical trial. Front Surg. 2023 Nov 10;10:1265370. doi: 10.3389/fsurg.2023.1265370. eCollection 2023. PMID 38026477